CLINICAL TRIAL: NCT03561363
Title: The Effect of 6 Weeks Saturated and Polyunsaturated High-Fat Diets on Insulin Sensitivity and Health Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Annemarie Lundsgaard, PostDoc. and principal investigator, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-3-2012-129
Record Dates: First submitted 2015-10-02; First posted 2018-06-19 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Insulin Sensitivity
Keywords: insulin sensitivity; high-fat diet
MeSH Terms: conditions — Insulin Resistance | interventions — Diet, High-Fat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Saturated high-fat diet (Experimental): In this intervention group, subjects ingest a saturated eucaloric high-fat diet (64 E%) with total fat content being similar to the polyunsaturated high-fat diet.
  The diet is enriched in saturated fat (36 E%). The main saturated fatty acids in the diet are primarily palmitic acid (C16:0) and stearic acid (C18:0). The main food sources are milk products, high-fat meat and vegetables.
  Carbohydrate comprise 20 E% and protein 15 E%.
  Interventions: Behavioral: High-fat diet
- polyunsaturated high-fat diet (Experimental): In this intervention group, subjects ingest a polyunsaturated eucaloric high-fat diet (64 E%), with total fat content being similar to the saturated high-fat diet. The diet is enriched in polyunsaturated fat (32 E%). The main polyunsaturated fatty acids in the diet are primarily linoleic acid (C18:2 n-6) and alpha-linoleic acid (C18:3 n-3). The main food sources are vegetable oils, nuts and high-fat fish (e.g. salmon). Carbohydrate comprise 20 E% and protein 15 E%.
  Interventions: Behavioral: High-fat diet

INTERVENTIONS:
Behavioral: High-fat diet — The aim of the intervention is to evaluate whether insulin sensitivity and selected Health parameters is affected, when the intake of saturated fatty acids or polyunsaturated fatty acids are highly increased, even when subjects are in energy balance.

SUMMARY:
The aim of the intervention is to gain insight into the long term effect of dietary fatty acid quality on insulin sensitivity and health parameters in healthy men.

Whole body and peripheral insulin sensitivity were measured, together with analyses of plasma hormones and metabolites. The plasma proteome was also analyzed. Molecular adaptations in skeletal muscle and adipose tissue were subject for investigation. Furthermore, gut microbiota population number and diversity will be analyzed from faeces samples obtained before and after the intervention.

DETAILED DESCRIPTION:
Two experimental diets with a high fat content (65 E% fat), enriched in either saturated or polyunsaturated fatty acids, were provided for 6 weeks to healthy men, in a randomized controlled intervention study with two arms.

Healthy, untrained, non-obese male subjects (27-45 years) were included in the study. The experimental diets are eucaloric, and thus provided so the subjects remains weight stable.

Before and after the intervention, two experimental days was conducted (2 experiments before and 2 experiments after the intervention).

At pre-intervention, subjects completed a high-fat meal test and insulin sensitivity was measured by the hyperinsulinemic-euglycemic clamp. On both days, blood and tissue biopsies were obtained. These two experimental days were repeated at the end of the 6 weeks intervention.

The hyperinsulinemic-euglycemic clamp was combined with stable isotope infusion (deuterium labelled glucose) in order to measure hepatic glucose production. Before the clamp, a catheter is inserted into the femoral vein, to enable measurement of insulin stimulated glucose uptake across the leg. Biopsies are obtained by the needle biopsy method from the vastus lateralis muscle and peri-umbilical subcutaneous adipose tissue. Blood samples were analyzed for glucose, insulin, inflammatory markers, gut hormones, adipokines, plasma fatty acid composition, and lipoprotein profile. Indirect calorimetric was also applied to measure substrate oxidation during the experimental days.

ELIGIBILITY:
Inclusion Criteria:

* healthy male subjects
* 27-45 years
* BMI 22-31
* maximal oxygen uptake <48 ml/kg/min

Exclusion Criteria:

* smokers
* use of medication
* parents with type-2 diabetes

Ages: 27 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change in whole body and peripheral insulin sensitivity | Each subject completes a hyperinsulinemic-euglycemic clamp at pre-intervention (week 0) and again after 6 weeks of intervention.
  This outcome will be evaluated with the hyperinsulinemic-euglycemic clamp, combined with the femoral arterio-venous balance technique

SECONDARY OUTCOMES:
Change in gut microbiota population number and diversity | Faeces samples are obtained from each subject at pre-intervention (week 0), and after the intervention (week 6). Analyses will be performed when the last faeces sample is obtained.
  Gut microbiota will be analyzed in faeces samples obtained from the subjects before and after the intervention (using 18s-RNA sequencing)

OTHER OUTCOMES:
Change in molecular adaptations in skeletal muscle and adipose tissue induced by saturated and polyunsaturated fatty acids | Biopsies are obtained at pre-intervention (week 0) and at week 6 after the intervention. Analyses will be performed when the last tissue biopsies are obtained.
  Skeletal muscle and subcutaneous adipose tissue biopsies are obtained from each subject. Specific molecular analyses (western blotting and real time-PCR) are applied to tissue samples to assess changes in relevant genes and proteins.

CONTACTS AND LOCATIONS:
Overall Officials: Bente Kiens, Professor, Principal Investigator — Dept. of Nutrition, Exercise and Sports, University of Copenhagen

REFERENCES:
- [Background] Vessby B, Uusitupa M, Hermansen K, Riccardi G, Rivellese AA, Tapsell LC, Nalsen C, Berglund L, Louheranta A, Rasmussen BM, Calvert GD, Maffetone A, Pedersen E, Gustafsson IB, Storlien LH; KANWU Study. Substituting dietary saturated for monounsaturated fat impairs insulin sensitivity in healthy men and women: The KANWU Study. Diabetologia. 2001 Mar;44(3):312-9. doi: 10.1007/s001250051620. PMID 11317662